CLINICAL TRIAL: NCT02325310
Title: Search for the Measles Vaccine Virus Excretion in Breast Milk of Breastfeeding Women After Postpartum Vaccination With a Combined Measles-mumps-rubella (MMR) Vaccine
Brief Title: Search for the Measles Vaccine Virus Excretion in Breast Milk of Breastfeeding Women After Postpartum Vaccination With MMR
Acronym: BREMEAVAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Service de Bactériologie-Virologie-Hygiène, CHU Limoge (Unknown); GO-CIC network (Réseau Gynéco-Obstetrical des Centres d'Investigation Clinique) (Unknown); REIVAC network (Réseau National d'Investigation Clinique en Vaccinologie) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-001538-28
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Measles; Rubella; Mumps
Keywords: Vaccine strain excretion in breast milk; Postpartum vaccination; Breastfeeding women; Measles-mumps-rubella vaccine; Breast milk; Vaccinology
MeSH Terms: conditions — Measles; Rubella; Mumps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breastfeeding women (Experimental): 70 breastfeeding women meeting all the inclusion criteria and none of the exclusion criteria will be immunized with MMR vaccine in postpartum (before the exit of the maternity)
  Interventions: Biological: Combined measles-mumps-rubella (MMR) vaccine - PRIORIX®

INTERVENTIONS:
Biological: Combined measles-mumps-rubella (MMR) vaccine - PRIORIX® — One dose of 0.5 mL vaccine will be administered (intra-muscularly or subcutaneous) in post-partum (before the exit of the maternity) during visit V0. A second dose will be administered at week 8(+/-15 days) during visit V1.

SUMMARY:
In order to assess the safety of breastfed infants after their mother's postpartum immunization with a combined measles-mumps-rubella (MMR) vaccine, the purpose of this study is to investigate whether measles vaccine strain is excreted in breast milk of breastfeeding women with negative rubella and measles serologies.

DETAILED DESCRIPTION:
This is a multicentre prospective study, to evaluate the safety of infant from 50 breastfeeding women, analyzable for primary endpoint, after postpartum immunization with MMR vaccine.

During the screening period, eligibility will be determined based on the inclusion and exclusion criteria. Medical records of pregnant women will be screened by study investigators, who will then propose to the woman to participate to the study during a phone call or a follow-up visit. Screening visit could take place 4 months before delivery planned date up until the day of delivery.

The investigator will explain the study to the woman. A copy of the informed consent documents will be given to the woman for reading and for further information about the study (by email, by post, or personally).

If the woman is willing to participate to the study and after she had given her screening informed consent, a blood sample for measles serological analysis will be drawn.

After signing the consent, women meeting all the inclusion criteria and none of the exclusion criteria will be vaccinated in post partum and before the exit of the maternity at day 0.

Each woman will have a blood draw at day 0 and breast milk samples as well as urine samples at the hospital at day 0 before vaccination.

Each included woman will also provide breast milk and urine home samples at days 7, 11 and 14 after vaccination. Reminder calls will be performed at days 7, 11 and 14 after vaccination.

Women will then be followed and vaccinated 8 weeks after the first vaccination, visit V1.

Each infant will be followed during 8 weeks. An optional blood sample for immunological analysis will be drawn at week 8 (visit v1). Informed consent form signed by the person(s) holding parental authority (both parents or mother only if the father has no parental authority) is needed for the infant to be included as well.

Diary cards will be used to follow the infant and the mother. If Infant and/or mother develop(s) suspected measles symptom(s), they will be evaluated by a study physician as soon as possible, preferably within 24 to 72 hours of acute measles symptom(s) onset.

In case of mother symptoms, infant will be also seen by a physician during mother's supplementary visit.

The visit at day 0 (V0) of the study will be performed at the maternity. The other visits, screening visit, V1 and supplementary visit (SV), will be performed either at the maternity or at the corresponding CIC if applicable. Home samples at 7, 11 and 14 days after vaccination will be directly sent at the laboratory of virology at Limoges. Home sampling can also be performed at the maternity or CIC according to their internal organization.

ELIGIBILITY:
Inclusion Criteria:

Women:

* Pregnant woman
* Age ≥ 18 years
* Planning to breastfeed her infant (mixed feeding is allowed)
* Having a negative serology for rubella during pregnancy
* Negative serology for measles based on the result from local laboratory
* Affiliated to a social security regimen

Infants:

* Informed consent form signed by the person(s) holding parental authority.
* Term newborn (≥36LMP)

Exclusion Criteria:

Women:

* Woman having a multiple pregnancy
* Woman planning to get pregnant in the month following the 2nd vaccination
* Woman with known or suspected HIV infection
* Woman with known or suspected immunodeficiency
* Woman with family history of hereditary immune deficiency
* Woman not mastering enough the reading / understanding of the French language to be able to consent to participate to the study
* Woman incapable to follow the procedures of the study and to respect study visits for the whole period of the study.
* Woman with contraindication for MMR vaccination:

  * Scarce hereditary problems of fructose intolerance
  * Woman with history of hypersensitivity to the active substances or to any of the excipients of the vaccine
  * Administration of human gammaglobulins in the past 3 to 11 months depending on the dose of human globulins administered (except for Rhophylac®)
  * Acute severe febrile illness within 7 days prior to injection
* Woman under systemic corticosteroids (prednisone, or equivalent ≥10 mg/day) within the previous 15 days or planning to use corticosteroids (i.e. prednisone, or equivalent ≥10 mg/day) during the 15 days following vaccination
* Woman under immunosuppressive therapy within the previous 3 months before vaccination or planning to use immunosuppressive therapy during the 15 days following vaccination Woman participating in any clinical trial with another investigational product 28 days prior to visit V0 or intent to participate in another clinical study with another investigational product at any time during the conduct of this study
* Any other reason which, according to the investigator, may interfere with the evaluation of the study objectives
* Woman with documented history of measles vaccination (1 or 2 doses) and/or history of documented measles

Infants:

* Blood draw is contraindicated or cannot be performed
* Infant with family history of hereditary immune deficiency
* Infant with suspected or confirmed immunodeficiency
* Any other reason which, according to the investigator, may interfere with the evaluation of the study objectives

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of the measles vaccine virus strain in breast milk. | day 7 after the first vaccination.
  Number of women with positive RT-PCR for measles vaccine virus strain in breast milk for at least one sample from day 7, 11 and 14 after postpartum vaccination with a combined measles-mumps-rubella (MMR) vaccine. RT PCR will be considered positive if the measurements exceed the limit of detection of 10 copies of genome per reaction
Prevalence of the measles vaccine virus strain in breast milk. | day 11 after the first vaccination.
  Number of women with positive RT-PCR for measles vaccine virus strain in breast milk for at least one sample from day 7, 11 and 14 after postpartum vaccination with a combined measles-mumps-rubella (MMR) vaccine. RT PCR will be considered positive if the measurements exceed the limit of detection of 10 copies of genome per reaction
Prevalence of the measles vaccine virus strain in breast milk. | day 14 after the first vaccination.
  Number of women with positive RT-PCR for measles vaccine virus strain in breast milk for at least one sample from day 7, 11 and 14 after postpartum vaccination with a combined measles-mumps-rubella (MMR) vaccine. RT PCR will be considered positive if the measurements exceed the limit of detection of 10 copies of genome per reaction

SECONDARY OUTCOMES:
Number of infants with reported clinical symptoms of measles | At V1 Visit (8 weeks +/- 15 days)
  Evaluation of the clinical impact of MMR vaccination in breastfeeding infant
Number of infants with reported clinical symptoms of measles | Between V0 visit and V1 visit (8 weeks +/- 15 days) after the first MMR vaccination
  Evaluation of the clinical impact of MMR vaccination in breastfeeding infant from data reported in the infant diary card (DiCa).
Number of women with reported clinical symptoms of measles | V1 Visit (8 weeks +/- 15 days) after the first MMR vaccination
  Evaluation of the clinical impact of MMR vaccination in breastfeeding infant from mother clinical data
Number of women with reported clinical symptoms of measles | Between V0 visit and V1 visit (8 weeks +/- 15 days) after the first MMR vaccination
  Evaluation of the clinical impact of MMR vaccination in breastfeeding infant from mother clinical data repoted in the diary card (DiCa).
Number of infants with positive measles serology (IgM) | V1 visit (8 weeks +/- 15 days) after the first MMR vaccination
  Evaluation of the immunological impact of MMR vaccination in breastfeeding infant.
Number of women with positive RT-PCR for measles vaccine virus strain in urine in at least one sample | At day 7 after the first vaccination.
  For detection of measles vaccine strain excretion in urine of breastfeeding women, the number of women, with negative rubella and measles serologies with positive RT-PCR for measles vaccine virus strain in urine for at least one sample from day 7, 11 and 14 after postpartum vaccination with a combined measles-mumps-rubella (MMR) vaccine will be assessed. RT PCR will be considered positive if the measurements exceed the limit of detection of 10 copies of genome per reaction
Number of women with positive RT-PCR for measles vaccine virus strain in urine in at least one sample | At day 11 after the first vaccination.
  For detection of measles vaccine strain excretion in urine of breastfeeding women, the number of women, with negative rubella and measles serologies with positive RT-PCR for measles vaccine virus strain in urine for at least one sample from day 7, 11 and 14 after postpartum vaccination with a combined measles-mumps-rubella (MMR) vaccine will be assessed. RT PCR will be considered positive if the measurements exceed the limit of detection of 10 copies of genome per reaction
Number of women with positive RT-PCR for measles vaccine virus strain in urine in at least one sample | At day 14 after the first vaccination.
  For detection of measles vaccine strain excretion in urine of breastfeeding women, the number of women, with negative rubella and measles serologies with positive RT-PCR for measles vaccine virus strain in urine for at least one sample from day 7, 11 and 14 after postpartum vaccination with a combined measles-mumps-rubella (MMR) vaccine will be assessed. RT PCR will be considered positive if the measurements exceed the limit of detection of 10 copies of genome per reaction
Quantification of the measles vaccine virus strain presented in breast milk in at least one sample | At day 7 after the first vaccination.
  In case of detection of measles vaccine virus strain excretion in breast milk, RT-PCR quantification measure of measles vaccine virus strain in woman breastmilk will be performed.
Quantification of the measles vaccine virus strain presented in breast milk in at least one sample | At day 11 after the first vaccination.
  In case of detection of measles vaccine virus strain excretion in breast milk, RT-PCR quantification measure of measles vaccine virus strain in woman breastmilk will be performed.
Quantification of the measles vaccine virus strain presented in breast milk in at least one sample | At day 14 after the first vaccination.
  In case of detection of measles vaccine virus strain excretion in breast milk, RT-PCR quantification measure of measles vaccine virus strain in woman breastmilk will be performed.
Microscopy assessment of the infectious activity of the measles vaccine virus presented in breast milk in at least one sample. | At day 7
  In case of detection of measles vaccine virus strain excretion in breast milk. The evaluation of the infectious activity of the measles vaccine virus will be performed using an in vitro infectivity assay. A result will be considered as positive when at least one positive fluorescent cell is detected.
Microscopy assessment of the infectious activity of the measles vaccine virus presented in breast milk in at least one sample. | At day 11 after the first vaccination.
  In case of detection of measles vaccine virus strain excretion in breast milk. The evaluation of the infectious activity of the measles vaccine virus will be performed using an in vitro infectivity assay. A result will be considered as positive when at least one positive fluorescent cell is detected.
Microscopy assessment of the infectious activity of the measles vaccine virus presented in breast milk in at least one sample. | At day 14 after the first vaccination.
  In case of detection of measles vaccine virus strain excretion in breast milk. The evaluation of the infectious activity of the measles vaccine virus will be performed using an in vitro infectivity assay. A result will be considered as positive when at least one positive fluorescent cell is detected.
Number of infant with positive salivary IgM/IgG | one year after the first vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Port Royal Hospital - Centre d'Investigation Clinique Cochin-Pasteur, Paris, France

REFERENCES:
- [Background] Alain S, Dommergues MA, Jacquard AC, Caulin E, Launay O. State of the art: Could nursing mothers be vaccinated with attenuated live virus vaccine? Vaccine. 2012 Jul 13;30(33):4921-6. doi: 10.1016/j.vaccine.2012.05.047. Epub 2012 May 31. PMID 22659446
- [Background] Chen LH, Zeind C, Mackell S, LaPointe T, Mutsch M, Wilson ME. Yellow fever virus transmission via breastfeeding: follow-up to the paper on breastfeeding travelers. J Travel Med. 2010 Jul-Aug;17(4):286-7. doi: 10.1111/j.1708-8305.2010.00430.x. No abstract available. PMID 20636609
- [Background] Losonsky GA, Fishaut JM, Strussenberg J, Ogra PL. Effect of immunization against rubella on lactation products. I. Development and characterization of specific immunologic reactivity in breast milk. J Infect Dis. 1982 May;145(5):654-60. doi: 10.1093/infdis/145.2.654. PMID 7077089
- [Background] Losonsky GA, Fishaut JM, Strussenberg J, Ogra PL. Effect of immunization against rubella on lactation products. II. Maternal-neonatal interactions. J Infect Dis. 1982 May;145(5):661-6. doi: 10.1093/infdis/145.2.661. PMID 7077090
- See also: Website of the CIC Cochin-Pasteur (CIC 1417) - 75679 Paris (France) — http://www.cicvaccinologie.com